CLINICAL TRIAL: NCT04277169
Title: A Volunteer Study to Collect Imaging Data for the Development of the IntelligentUltrasound Anatomy Guide
Status: Completed | Type: Observational
Sponsor: IntelligentUltrasound Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: IU2020_AG_04
Record Dates: First submitted 2020-01-23; First posted 2020-02-20 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Ultrasound Imaging of Anatomical Structures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a single-centre, prospective, non-randomised volunteer study to be undertaken in the MediCentre, Heath Park, Cardiff, UK

DETAILED DESCRIPTION:
This is a single-centre, non-randomised, prospective study involving at least 120 participants. The data collected in this study will augment the data collected in IU2019_AG_03 Volunteers will be enrolled sequentially until at least 120 scans have been recorded. Ideally, between 120 and 150 scans will be recorded.

Phase I Data collected from up to the first 80 participants in each of the six peripheral nerve block areas will be used as a training/verification set. This set will be used to develop and verify models for the identification and highlighting of target anatomical structures on ultrasound images.

Phase II The remaining 40 videos in each area (total minimum 120 participants) will be used for validation of these models.

The validation videos will be fed into the models created during Phase I of the study and the output anatomy highlighting will be recorded as a separate video, overlaid on the original ultrasound image. The overlay video will then be further split into 30-second segments.

A panel of three independent expert anaesthetists will be convened to review and score the segments for accuracy and performance to the endpoints agreed in Phase I of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 18 years of age;
2. Able to comprehend and sign the Informed Consent prior to enrolment in the study.

Exclusion Criteria:

1. Aged <18 years of age;
2. Unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers who respond to adverts placed at the University Hospital of Wales (UHW) and related sites in Cardiff.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Model development and verification | 4 months
  Collection of ultrasound scans. The collected scans will be assessed and used in the development and verification of deep-learning models that identify the target structures using a training dataset.

SECONDARY OUTCOMES:
Model validation | 4 months
  Estimation of performance and accuracy (e.g. success/failure of highlighting of target structures, average distance of highlighting from target, time spent highlighting correct structure as a proportion of time target visible)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Margetts, Study Director — IntelligentUltrasound Limited
Locations (1):
- MediCentre, Heath Park, Cardiff, Wales, United Kingdom